CLINICAL TRIAL: NCT01158651
Title: A Phase II Study of RAD001 (Everolimus) for Children With NeurF1 and Chemotherapy-Refractory Radiographic Progressive Low Grade Gliomas
Brief Title: Everolimus for Children With NF1 Chemotherapy-Refractory Radiographic Progressive Low Grade Gliomas
Acronym: NFC-RAD001
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Boston Children's Hospital (Other); Children's Hospital of Philadelphia (Other); Children's National Research Institute (Other); Children's Hospital Medical Center, Cincinnati (Other); National Cancer Institute (NCI) (NIH); University of Chicago (Other); University of Utah (Other); Washington University School of Medicine (Other); Ann & Robert H Lurie Children's Hospital of Chicago (Other); NYU Langone Health (Other); Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, Bruce Korf, MD, Principal Investigator, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: DOD W81XWH-05-1-0615; UAB (Other Grant/Funding Number: UAB F100225004); NCT00652990 (obsolete NCT alias)
Record Dates: First submitted 2010-07-02; First posted 2010-07-08 (Estimated); Results first posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Glioma
Keywords: NF1; low-grade glioma; progressive; children; NF Type 1 - low grade glioma - not responded to treatments
MeSH Terms: conditions — Glioma | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- RAD001 (Everolimus) Active Therapy (Experimental): If you take part in this research study, you will be given a participant diary for each treatment course to help you keep track of when you take your RAD001. You will be required to bring the completed diary at each scheduled visit. A treatment "course" lasts 4 weeks and there will not be any breaks between courses. You may stay on study for a total of 12 courses (48 weeks).
  You will take the study medication (tablets) by mouth, once a day during each course for as long as you are participating in this study. You will also be required to take an antibiotic during treatment to prevent infection.
  Interventions: Drug: RAD001 (Everolimus)

INTERVENTIONS:
Drug: RAD001 (Everolimus) — If you take part in this research study, you will be given a participant diary for each treatment course to help you keep track of when you take your RAD001. You will be required to bring the completed diary at each scheduled visit. A treatment "course" lasts 4 weeks and there will not be any breaks between courses. You may stay on study for a total of 12 courses (48 weeks).
  You will take the study medication (tablets) by mouth, once a day during each course for as long as you are participating in this study. You will also be required to take an antibiotic during treatment to prevent infection.
  Other Names: RAD001; Everolimus

SUMMARY:
The purpose of this research study is to learn if the study drug RAD001 can shrink or slow the growth of low-grade gliomas in children with Neurofibromatosis type 1 (NF1). Additionally, the safety of RAD001 will be studied.

The study drug, RAD001, is a drug that may act directly on tumor cells by preventing tumor cell growth and development. RAD001 has been studied in participants with various types of cancer as a single agent (a drug that is used alone to treat the cancer) or in combination with a number of well known anticancer therapies. Information from these research studies suggests that RAD001 may help to shrink or slow the growth of low-grade gliomas.

In this research study, the investigators are looking to see the response of RAD001 in children with low-grade gliomas and NF1 that have either not responded to treatment or have come back after treatment. We are also looking for the highest dose of RAD001 that can be given safely in this patient population.

DETAILED DESCRIPTION:
After signing this consent form, you will be asked to undergo some screening tests or procedures to find out if you can be in the research study. These tests and procedures are likely to be part of regular glioma care and may be done even if it turns out that you do not take part in the research study. If you have had some of these tests or procedures recently, they may or may not have to be repeated.

A medical history, which involves questions about your health history, any medications you are taking or plan to take, and any allergies.

A physical exam, during which you will be asked about any problems that you might be having. Additionally, your clinician will check your vital signs (body temperature, heart rate, breathing rate, and blood pressure) and bodily systems (respiratory, nervous, digestive, etc). The doctor will also evaluate your performance status, which indicates how much your illness affects your activity level.

Blood tests, including tests to measure any effects of your disease. Approximately 1-2 teaspoons of blood will be drawn for these tests.

Urine test, which will be done to make sure your kidneys are functioning properly.

An assessment of your tumor using scans of the brain. MRI (Magnetic Resonance Imaging) will be used to look at and evaluate the tumor.

An Electrocardiogram (ECG), which measures the electrical activity of your heart

A pregnancy test for females of childbearing potential. A small amount of blood (about half a teaspoon) or urine will be drawn for this test.

If these tests show that you are eligible to participate in the research study, you will begin the study treatment. If you do not meet the eligibility criteria, you will not be able to participate in this research study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis: All patients must have a radiographically progressive low-grade glioma and at least two of the following diagnostic criteria for NF1, and/or a pathogenic NF1 gene mutation demonstrated in peripheral blood-derived DNA:
* Six or more café-au-lait spots (greater than or equal to 0.5 cm in prepubertal subjects or greater than or equal to 1.5 cm in postpubertal subjects)
* Freckling in the axilla and/or inguinal region
* Plexiform neurofibroma
* Two or more Lisch nodules
* A distinctive bony lesion (dysplasia of the sphenoid bone or dysplasia or thinning of long bone cortex)
* A first-degree relative with NF1
* An optic pathway glioma
* Disease Status: All patients must have radiographically progressive low-grade glioma (including NF1 related visual pathway gliomas) after failure of a carboplatin-containing regimen. Patients with recurrent/progressive disease do not require a biopsy to confirm the diagnosis.
* Evaluable or Measurable Disease: Patients must have at least one evaluable or measurable site of disease according to criteria described in Section 9. If the patient has had previous radiation to the marker lesion(s), there must be evidence of progression since the radiation.
* Age: Patients must be greater than 1 years and less than or equal to 21 years of age at the time of study entry.
* Performance Level: Karnofsky 50% for patients greater than 10 years of age and Lansky 50% for patients 10 years of age (Appendix I). Note: Patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.
* Prior Therapy
* Patients must have failed or not been able to tolerate a carboplatin-based regimen.
* Patients must have fully recovered from the acute toxic effects of all prior chemotherapy or radiotherapy prior to entering this study.
* Myelosuppressive chemotherapy: Must not have received within 4 weeks of entry onto this study (6 weeks if prior nitrosourea).
* Hematopoietic growth factors: At least 7 days since the completion of therapy with a growth factor.
* Biologic (anti-neoplastic agent): At least 14 days since the completion of therapy with a biologic agent. For agents that have known adverse events occurring beyond 14 days after administration, this period must be extended beyond the time during which adverse events are known to occur. These patients must be discussed with the Study Chair on a case-by-case basis.
* Investigational Drugs: Patients must not have received an investigational drug within 14 days.
* Steroids: Patients with endocrine deficiencies are allowed to receive physiologic or stress doses of steroids if necessary.
* Cytochrome P450 3A4 (CYP3A4) inhibitors: Patients may not be currently receiving strong inhibitors of CYP3A4, and may not have received these medications within 1 week prior to study entry. These include:
* Antibiotics: clarithromycin, erythromycin, troleandomycin Anti-HIV agents: delavirdine, nelfinavir, amprenavir, ritonavir, indinavir, saquinavir, lopinavir
* Antifungals: itraconazole, ketoconazole, fluconazole (doses greater than 200 mg/day), voriconazole
* Antidepressants: nefazodone, fluvoxamine Calcium channel blockers: verapamil, diltiazem
* Miscellaneous: amiodarone,
* In addition, grapefruit juice should be avoided, as it inhibits CYP3A4.
* CYP3A4 inducers: Patients must also avoid St. John's Wort, an inducer of CYP3A4
* Enzyme inducing anticonvulsants: Patients may not be taking enzyme-inducing anticonvulsants, and may not have received these medications within 1 week prior to study entry, as these patients may experience different drug disposition. These medications include:
* Carbamazepine (Tegretol)
* Felbamate (Felbatol)
* Phenobarbitol
* Phenytoin (Dilantin)
* Primidone (Mysoline)
* Oxcarbazepine (Trileptal)
* Radiation therapy (XRT):
* 6 months must have elapsed if the patient has received involved field XRT or gamma knife that includes all target lesions (i.e., there is no restriction if a new lesion arises outside the radiation field or a non-irradiated lesion progresses);
* 6 months must have elapsed if the patient has received craniospinal XRT.
* 6 weeks must have elapsed if patient has received radiation to areas outside optic glioma.
* Surgery: At least 2 weeks must have elapsed since undergoing major surgery.
* Organ Function Requirements:
* Adequate Bone Marrow Function Defined as:

  * Peripheral absolute neutrophil count (ANC) __1000/__L
  * Platelet count __ 100,000/__ L (transfusion independent)
  * Hemoglobin __ 9.0 gm/dL (may receive red blood cell (RBC) transfusions)
* Adequate Renal Function Defined As:

  - A serum creatinine based on age as follows: Age (Years) Maximum Serum Creatinine (mg/dL)

  __5 / 5 less than age __ 10 / 10 less than age __ 15/ greater than 15 0.8 1.0 1.2 1.5 OR a creatinine clearance or radioisotope glomerular filtration rate (GFR) __ 70ml/min/1.73 m2
* Adequate Liver Function Defined As:

  * Bilirubin (sum of conjugated + unconjugated) __ 1.5 x upper limit of normal (ULN) for age, and
  * Serum glutamic pyruvic transaminase (SGPT) (alanine transaminase (ALT)) __ 5 x upper limit of normal (ULN) for age, and
  * Serum albumin __ 2 g/dL
  * International normalised ratio (INR) less than 1.3 (or less than 3 on anticoagulants)
  * Serum creatinine less than or equal to 1.5x ULN
* Fasting Low-density lipoprotein cholesterol (LDL) Cholesterol:

  * Patients must have a fasting LDL cholesterol within the normal range per institutional guidelines
  * Patients taking a cholesterol lowering agent must be on a single medication and on a stable dose for at least 4 weeks
* Fasting Serum Cholesterol:

  - less than or equal to 300 mg/dL OR less than or equal to 7.75 mmol/L AND fasting triglycerides less than or equal to 2.5x ULN. NOTE: In case one or both of these thresholds are exceeded, the patient can only be included after initiation of appropriate lipid lowering medication.
* Signed informed consent/assent

Exclusion Criteria:

* Chronic treatment with systemic steroids or another immunosuppressive agent. Patients with endocrine deficiencies are allowed to receive physiologic or stress doses of steroids if necessary.
* Evidence of an active lesion including: plexiform neurofibroma, malignant peripheral nerve sheath tumor, or other cancer requiring concurrent treatment with chemotherapy or radiation therapy. Patients not requiring treatment for these lesions are eligible for this protocol.
* Patients who:

  * have had a major surgery or significant traumatic injury within 2 weeks of start of study drug;
  * have not recovered from the side effects of any major surgery (defined as requiring general anesthesia but excluding a procedure for insertion of central venous access), or
  * may require major surgery during the course of the study.
* Other malignancies within the past 3 years except for adequately treated carcinoma of the cervix or basal or squamous cell carcinomas of the skin.
* Uncontrolled brain or leptomeningeal metastases, including patients who continue to require glucocorticoids for brain or leptomeningeal metastases.
* Patients with an active, bleeding diathesis or on oral anti-vitamin K medication (except low dose coumarin).
* Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study such as:

  * symptomatic congestive heart failure of New York heart Association Class III or IV.
  * unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction within 6 months of start of study drug, serious uncontrolled cardiac arrhythmia or any other clinically significant cardiac disease.
  * severely impaired lung function.
  * uncontrolled diabetes as defined by fasting serum glucose greater than 1.5x ULN.
  * active (acute or chronic) or uncontrolled severe infections.
  * liver disease such as cirrhosis, chronic active hepatitis or chronic persistent hepatitis.
* Other concurrent severe and/or uncontrolled medical disease which could compromise participation in the study (i.e., uncontrolled diabetes, uncontrolled hypertension, severe infection, severe malnutrition, chronic liver or renal disease, active upper gastrointestinal (GI) tract ulceration).
* A known history of HIV seropositivity or known immunodeficiency.
* Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of RAD001 (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or small bowel resection). A nasogastric tube (NG tube) is allowed.
* Women who are pregnant or breast feeding.
* Males or females of reproductive potential may not participate unless they have agreed to use an effective contraceptive method during the time they are receiving the study drug and for 3 months thereafter. Abstinence is an acceptable method of birth control. Oral, implantable, or injectable contraceptives may be affected by cytochrome P450 interactions, and are therefore not considered effective for this study. Women of childbearing potential will be given a pregnancy test within 7 days prior to administration of RAD001 and must have a negative urine or serum pregnancy test.
* Patients who have received prior treatment with a mammalian target of rapamycin (mTOR) inhibitor.
* Dental braces or prosthesis that interferes with tumor imaging.
* History of noncompliance to medical regimens.
* Patients unwilling to or unable to comply with the protocol or who, in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study.

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 23 (Actual)
Dates: Start 2010-07-10 (Actual); Primary Completion 2014-09-04 (Actual); Study Completion 2017-10-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce R. Korf, MD, PhD, Study Chair — The University of Alabama at Birmingham; Mark Kieran, MD, Principal Investigator — Boston Children's Hospital
Locations (12):
- United States (12):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Lurie Hospital, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - National Cancer Institute, Bethesda, Maryland
  - Children's Hospital Boston, Boston, Massachusetts
  - Washington University, St Louis, Missouri
  - New York University Medical Center, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Utah, Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Groups:
- RAD001 (Everolimus) Active Therapy: If you take part in this research study, you will be given a participant diary for each treatment course to help you keep track of when you take your RAD001. You will be required to bring the completed diary at each scheduled visit. A treatment "course" lasts 4 weeks and there will not be any breaks between courses. You may stay on study for a total of 12 courses (48 weeks).
  You will take the study medication (tablets) by mouth, once a day during each course for as long as you are participating in this study. You will also be required to take an antibiotic during treatment to prevent infection.
  RAD001 (Everolimus): If you take part in this research study, you will be given a participant diary for each treatment course to help you keep track of when you take your RAD001. You will be required to bring the completed diary at each scheduled visit. A treatment "course" lasts 4 weeks and there will not be any breaks between courses. You may stay on study for a total of 12 course
Period: Overall Study
Arm/Group | RAD001 (Everolimus) Active Therapy
Started | 23
Completed | 22
Not Completed | 1

BASELINE CHARACTERISTICS:
Groups:
- Active Therapy: If you take part in this research study, you will be given a participant diary for each treatment course to help you keep track of when you take your RAD001. You will be required to bring the completed diary at each scheduled visit. A treatment "course" lasts 4 weeks and there will not be any breaks between courses. You may stay on study for a total of 12 courses (48 weeks). You will take the study medication (tablets) by mouth, once a day during each course for as long as you are participating in this study. You will also be required to take an antibiotic during treatment to prevent infection. If you take part in this research study, you will be given a participant diary for each treatment course to help you keep track of when you take your RAD001. You will be required to bring the completed diary at each scheduled visit. A treatment "course" lasts 4 weeks and there will not be any breaks between courses. You may stay on study for a total of 12 courses (48 weeks).
Arm/Group | Active Therapy
Number analyzed (Participants) | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.8 (4.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 21
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 21
  More than one race | 0
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: RAD001 Response Rate Based on 2D MRI Change From Baseline
Description: Outcome is 2D MRI target tumor volume compared to baseline volume. Success criteria is volume less than 80% of baseline.
Time Frame: Approximately 48 weeks
Population: Intent to treat
Measure: Number (95% Confidence Interval); unit: participants
Groups:
- RAD001 (Everolimus) Active Therapy: If you take part in this research study, you will be given a participant diary for each treatment course to help you keep track of when you take your RAD001. You will be required to bring the completed diary at each scheduled visit. A treatment "course" lasts 4 weeks and there will not be any breaks between courses. You may stay on study for a total of 12 courses (48 weeks). You will take the study medication (tablets) by mouth, once a day during each course for as long as you are participating in this study. You will also be required to take an antibiotic during treatment to prevent infection. If you take part in this research study, you will be given a participant diary for each treatment course to help you keep track of when you take your RAD001. You will be required to bring the completed diary at each scheduled visit. A treatment "course" lasts 4 weeks and there will not be any breaks between courses. You may stay on study for a total of 12 courses (48 weeks).
Arm/Group | RAD001 (Everolimus) Active Therapy
Number analyzed (Participants) | 22
participants | 15 [11 to 19]
Statistical Analysis 1: Comparison: RAD001 (Everolimus) Active Therapy; Test type: Superiority — The treatment regimen was considered promising for further study if after 48 weeks of treatment there was at least a 25% response rate compared to an expected response rate of 5% or less, which was considered evidence of an unpromising regimen. Assuming the true response rate is 5%, the binomial distribution was used to calculate Type I errors and power; p < 0.001, Exact test; Proportion responding = 0.682, 95% CI 2-sided [0.4872 to 0.8764]

2. Secondary Outcome: Common Terminology Criteria for Adverse Events (CTCAE) Events
Description: Number of participants experiencing serious CTCAE events in the study.
Time Frame: approximately 48 weeks
Measure: Number; unit: participants
Arm/Group | RAD001 (Everolimus) Active Therapy
Number analyzed (Participants) | 23
participants | 23

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | RAD001 (Everolimus) Active Therapy
All-Cause Mortality (participants affected / at risk) | 1/23
Serious Adverse Events (participants affected / at risk) | 6/23
Other Adverse Events (participants affected / at risk) | 21/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RAD001 (Everolimus) Active Therapy (N=23)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Cardio Respiratory Arrest (Cardiac disorders) | 1 (1)
Dehydration (Gastrointestinal disorders) | 1 (1)
Diabetes insipidus (Endocrine disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Electrolyte disturbance (Investigations) | 1 (1)
Hydrocephalus (Nervous system disorders) | 1 (1)
Hypernatremia (Investigations) | 1 (1)
Hypokalemia (Investigations) | 1 (1)
Infection with absolute neutrophil count (ANC) (Infections and infestations) | 1 (1)
Low hemoglobin (Blood and lymphatic system disorders) | 1 (1)
Pelvic Mass (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Shunt Malfunction (Nervous system disorders) | 1 (1)
Resection of right temporal lobe tumor (Surgical and medical procedures) | 1 (1)
Blindness (Eye disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
brain surgery (Surgical and medical procedures) | 1 (1)
Brain resection (Surgical and medical procedures) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RAD001 (Everolimus) Active Therapy (N=23)
Leukopenia (Blood and lymphatic system disorders) | 4 (4)
Neutropenia (Blood and lymphatic system disorders) | 4 (4)
Hyperlipidemia (Metabolism and nutrition disorders) | 2 (2)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 2 (2)
Mucositis (Gastrointestinal disorders) | 9 (9)
Other non-hematologic toxicity (Investigations) | 10 (36)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No